CLINICAL TRIAL: NCT04149041
Title: The Applications of Point-of-care Ultrasound in ED Unselected, Non-critical Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201907173RIND
Record Dates: First submitted 2019-10-24; First posted 2019-11-04 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2019-10

CONDITIONS: Ultrasound Therapy; Complications
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound — POCUS is applied to adult patients in an emergency department.

SUMMARY:
to investigate prevalence of agreement between sonographic and clinical diagnosis in adult patients seen in an emergency department.

DETAILED DESCRIPTION:
Point-of-care ultrasound (POCUS) can improve patient management in the emergency department (ED). However, previous studies have focused only on selected groups of patients, such as trauma, shock, dyspnea, or critically ill patients, or patients with an already known diagnosis. Most patients seen in the ED do not match these criteria. This study aims to investigate prevalence of agreement between sonographic and clinical diagnosis in adult patients seen in an emergency department.

ELIGIBILITY:
Inclusion Criteria:

* adult patients in the emergency department receiving ultrasonographic examinations were enrolled.

Exclusion Criteria:

* adult patients in the emergency department not receiving ultrasonographic examinations.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From June 2014 to August 2019, adult patients in the emergency department receiving ultrasound were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
number of agreement between the sonographic diagnosis and the clinical diagnosis | one month
  ultrasound
length of stay at the emergency department | one month
  length of stay

CONTACTS AND LOCATIONS:
Overall Officials: National Taiwan University Hospital, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang CT, Wang LW, Lin SY, Chen TY, Ho YJ, Wang PH, Liu KL, Wu YM, Wang HP, Lien WC. Impact of a POCUS-first versus CT-first approach on emergency department length of stay and time to surgical consultation in patients with acute cholecystitis: a retrospective study. Scand J Trauma Resusc Emerg Med. 2025 Feb 10;33(1):28. doi: 10.1186/s13049-025-01341-2. PMID 39930510
- [Derived] Wang PH, Chen JY, Ling DA, Lee AF, Ko YC, Lien WC, Huang CH. Earlier point-of-care ultrasound, shorter length of stay in patients with acute flank pain. Scand J Trauma Resusc Emerg Med. 2022 Apr 21;30(1):29. doi: 10.1186/s13049-022-01017-1. PMID 35449010